CLINICAL TRIAL: NCT07208253
Title: Effect of Dexamethasone and Bupivacaine on Postoperative Pain Following Total Extraperitoneal Hernioplasty: A Randomized Controlled Prospective Study
Brief Title: Dexamethasone and Bupivacaine for Pain After Hernia Surgery
Acronym: DEXA-BUPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gürkan Değirmencioğlu (Other Government)
Responsible Party: Sponsor-Investigator, Gürkan Değirmencioğlu, General Surgery Specialist, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EŞH-GC-2025-01; 2021/26 (Other: Mustafa Kemal University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Inguinal Hernia Repair (Not Urgent)
Keywords: Inguinal Hernia, Total Extraperitoneal Hernioplasty (TEP), Postoperative Pain, Dexamethasone, Bupivacaine, Randomized Controlled Trial
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, parallel assignment study comparing dexamethasone plus bupivacaine versus no local treatment in patients undergoing elective unilateral laparoscopic total extraperitoneal (TEP) hernioplasty.
Who Masked: Outcomes Assessor
Masking Description: Pain scores were assessed by an independent health care provider who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Patients received 20 mg bupivacaine (4 mL of 0.5%) combined with 8 mg dexamethasone. The solution was sprayed over the mesh and surrounding tissues after mesh placement during laparoscopic total extraperitoneal (TEP) hernioplasty.
  Interventions: Drug: Bupivacaine + Dexamethasone
- No Intervention: Control Group (No Intervention): Patients underwent standard laparoscopic total extraperitoneal (TEP) hernioplasty without local application of bupivacaine or dexamethasone in the operative field.

INTERVENTIONS:
Drug: Bupivacaine + Dexamethasone — 20 mg bupivacaine (4 mL of 0.5%) combined with 8 mg dexamethasone, sprayed locally over the mesh and surrounding tissues after placement during laparoscopic TEP hernioplasty.
  Arms: Experimental: Intervention Group

SUMMARY:
This study looked at whether a combination of two medicines, dexamethasone and bupivacaine, can reduce pain after laparoscopic hernia surgery. A total of 175 patients who had elective total extraperitoneal (TEP) hernia repair were randomly assigned to two groups. One group received a spray of dexamethasone and bupivacaine around the surgical mesh, while the other group did not receive any local treatment.

Pain levels were measured at 3, 6, and 12 hours after surgery using a visual pain scale. The need for additional pain medicine and patient satisfaction were also recorded. Patients who received dexamethasone and bupivacaine reported lower pain scores, needed less extra pain medicine, and were more satisfied with their pain control compared to the control group.

The results suggest that this simple, safe, and low-cost method may help improve pain control and comfort after laparoscopic hernia repair.

DETAILED DESCRIPTION:
This randomized controlled study investigated the effect of adding dexamethasone to bupivacaine for pain management after laparoscopic total extraperitoneal (TEP) hernia repair. Postoperative pain is still a significant concern after TEP, even though this minimally invasive technique generally causes less pain than open surgery. Local anesthetics such as bupivacaine are widely used, but their effect is limited in duration. Dexamethasone, an anti-inflammatory corticosteroid, has been shown to enhance and prolong analgesia when combined with local anesthetics.

A total of 175 patients undergoing elective unilateral TEP hernioplasty were randomized into two groups. The intervention group received 20 mg of bupivacaine (4 mL of 0.5%) mixed with 8 mg dexamethasone, sprayed directly on the surgical mesh and surrounding tissues after mesh placement. The control group did not receive any local treatment in the operative field. All patients received standard postoperative analgesia.

Pain scores were assessed using the Visual Analog Scale (VAS) at 3, 6, and 12 hours after surgery. The need for additional analgesics, patient satisfaction, and early complications were also recorded.

Results showed that patients in the dexamethasone + bupivacaine group had significantly lower pain scores at all time points, required fewer additional analgesics, and reported higher satisfaction compared to controls. No increase in surgical complications was observed.

This study suggests that the local application of dexamethasone combined with bupivacaine is a safe, simple, and cost-effective method to improve early postoperative pain control and patient comfort after laparoscopic TEP hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) scheduled for elective unilateral inguinal hernia repair with the laparoscopic total extraperitoneal (TEP) technique
* American Society of Anesthesiologists (ASA) physical status I-II
* Ability to provide informed consent

Exclusion Criteria:

* Age <18 years
* ASA physical status ≥III
* Recurrent or bilateral inguinal hernia
* History of allergy to local anesthetics or corticosteroids
* Chronic opioid use or dependence
* Severe hepatic, renal, or cardiac disease
* Pregnancy or breastfeeding
* Patients who declined to participate or could not provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores | 12 hours after surgery
  Pain intensity measured using the Visual Analog Scale (VAS) at 3, 6, and 12 hours after surgery.

SECONDARY OUTCOMES:
Additional Analgesic Requirement | 24 hours after surgery
  Number of patients requiring supplemental analgesics during the first 24 hours after surgery.
Patient Satisfaction | Within 24 hours after surgery
  Patient-reported satisfaction with pain management, scored on a 4-point Likert scale (poor, moderate, good, excellent).
Postoperative Complications | Within 30 days after surgery
  Frequency of early complications such as hematoma, urinary retention, wound infection.

CONTACTS AND LOCATIONS:
Overall Officials: GÜRKAN DEĞİRMENCİOĞLU, MD, Principal Investigator — Etlik City Hospital, Department of General Surgery, Ankara,Turkey
Locations (1):
- Etlik City Hospital (Etlik Şehir Hastanesi), Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because this was a single-center study with a limited sample size, and data sharing is not planned in the study protocol.